CLINICAL TRIAL: NCT04259957
Title: How do Staff Experience Incorporating Immersive Virtual Reality in a Chronic Pain Management Group: a Qualitative Assessment
Brief Title: Staff Experiences of Using Virtual Reality in a Pain Management Group
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: InHealth Group (Industry)
Responsible Party: Principal Investigator, Thomas Shelton, Clinical Lead, InHealth Group
Other Study IDs: 01
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain
Keywords: Virtual Reality
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinician using Virtual Reality in Pain Management Program: Clinicians who have used immersive virtual reality as part of Pain Management program group.
  Interventions: Device: Immersive Virtual Reality

INTERVENTIONS:
Device: Immersive Virtual Reality — Immersive virtual reality games and mindfulness in Oculus Quest Virtual Reality headset

SUMMARY:
Immersive Virtual Reality is a fast developing technology that allows a number of opportunities to engage people in activities that they otherwise might find difficult. For instance exercising in a fun way when they have difficulty exercising in the way they previously enjoyed. Alternatively the immersive nature of the experience might make it easier to engage in tasks in an otherwise distracting world.

The investigators are interested in exploring how Virtual Reality games and programs can help people with Chronic Pain. Working with Researchers at Sheffield Hallam University the research team introduced Virtual Reality headsets and games to people engaging in a Pain Management Program Group lasting 6 weeks for 3 hours a week. This involved NHS patients in the UK, delivered by a physiotherapist and an occupational therapist. This group involved 8 individuals with a variety of chronic pain conditions. Patients used Virtual Reality headsets and games throughout the program to aid exercise and mindfulness activities.

This is a relatively new approach and the investigators are not aware of any other organisations making use of this technology in this way. It would be useful developing its use to explore the issues those leading the Pain Management Group and supporting patients found. Speaking to these individuals in interviews will explore their experiences and feelings deeply and allow us to learn about what worked well and what challenges they faced. These interviews would be conducted in a format of qualitative research that would explore the experiences staff had, and compare it to other experiences of introducing patient-used technology in healthcare.

DETAILED DESCRIPTION:
This is a new technology and form of clinical treatment. As such it is not possible to draw on existing literature to give a hypothesis. Rather this research will aim to help form new understanding of this developing technological approach. Subsequently a qualitative approach is best to gain an indepth and detailed understanding of the experiences of the clincians who delivered Virtual Reality in a chronic pain group structure. In the group, around 8 patients with Chronic, non-cancer pain were given the opportunity to use a range of programs; demos for commercially available computer games, a virtual natural world to support use of mindfulness approaches, and a program developed for us by Sheffield Hallam University involving climbing and bow and arrow components.

Individual semi-structured interviews will allow the researchers to focus on aspects of the delivery of the technology and how it might be improved in the future. It will also give the freedom to respond to the participating clinicians and explore previously unanticipated issues or views.

The Pain Management Program Group runs over 6 weeks. Exercise components and mindfulness makes up part of each session and is normally led by the clinician. They are largely made up of educational components that will be led as normal. In these Virtual Reality Pain Management Groups the exercise component will be replaced by active games in a virtual reality environment. This will involve a range of games that engage the patient to move their upper-limbs and trunk. The mindfulness component will place the patient in the immersive digital environment and then encourage them to engage with it by making use of conventional mindfulness exercises.

At a date following the completion of the group, the staff leading the group will be involved in a single semi-structured interview lasting around 30 minutes. Participants will be asked about how they found using Virtual Reality technology in a Pain Management Group, what issues arose that they had to overcome and how they think the sessions need to be developed in the future. Interviews will take place during clinic times over the telephone. Time will be allowed so that staff can take part in these interviews. The interviewer will be another member of staff at the same organisation who has not been involved in the delivery of the Virtual Reality technology. They are also the chief investigator.

The interviews will be recorded directly onto a secure laptop (password protected encryption) and the recordings will be stored on a secure server in a password protected file. It will be transcribed and analysed in Microsoft Word using a thematic approach. This will then be transferred to the Sheffield Hallam University Data Archive following analysis.

Confirmation of the themes identified and outcomes of the qualitative research will be reviewed with the interviewed clinicians. This will attempt to address researcher bias and ensure that participants recognise the issues raised by the research.

ELIGIBILITY:
Inclusion Criteria:

* Must be a qualified health care professional. Must work for Inhealth Pain Management in the West Lancashire team. As part of the above treating those with chronic (longer than 3 months) non-cancer pain.

Must have delivered at lest one session of the Pain Management Program with use of Immersive Virtual Reality.

Exclusion Criteria:

* Any clinician who is voluntarily unwilling to take part in the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinicians working at INHEALTH Pain Management in the West Lancashire CCG area, UK.
  Clinicians who have worked with patients in the Pain Management Program group using virtual reality.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview Qualitative interview | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Inhealth Pain Management, Barnsley, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No